CLINICAL TRIAL: NCT03048474
Title: Ipilimumab and Nivolumab in the Treatment of Malignant Pleural Mesothelioma: a Phase II Study. Acronym: INITIATE
Brief Title: Ipilimumab and Nivolumab in the Treatment of Malignant Pleural Mesothelioma
Acronym: INITIATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16INM
Record Dates: First submitted 2016-10-24; First posted 2017-02-09 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: progressive disease after at least 1 course of chemotherapy
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab and Ipilimumab (Experimental): Nivolumab will be administered at a fixed dose of 240 mg every 2 weeks for a maximum period of 2 years. Nivolumab will be given in combination with ipilimumab on week 1, 7, 13 and 19. Ipilimumab will be administered at the dose of 1 mg/Kg.
  Interventions: Drug: nivolumab and ipilimumab

INTERVENTIONS:
Drug: nivolumab and ipilimumab
  Other Names: BMS-936558 and L01XC11

SUMMARY:
This is a prospective, monocenter, single arm, phase II trial in 33 patients with unresectable MPM, who experience disease progression or recurrence after at least one previous line of platinum-based systemic treatment.

Nivolumab will be administered at a fixed dose of 240 mg every 2 week. Nivolumab will be given in combination with ipilimumab on week 1, 7, 13 and 19 and will be administered prior to the infusion of ipilimumab. Ipilimumab will be administered at the dose of 1 mg/Kg.The patients will receive nivolumab monotherapy on week 3, 5, 9, 11, 15 and 17. From week 21 thereafter, Nivolumab will be then administered every 2 weeks for a maximum period of 2 years or until disease progression or unacceptable toxicity occurs.

DETAILED DESCRIPTION:
Patients will undergo pre- and post-treatment thoracoscopies/biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥ 18 years
* WHO-ECOG performance status 0 or 1
* Able to comply with the study protocol, in the investigator's judgment
* Patients with histologically confirmed diagnosis of the recurrence of MPM. Any pleural MPM subtype is permitted for inclusion in the study
* Progressive disease after at least one prior systemic treatment with a platinum-based doublet (both cisplatin and carboplatin are allowed) for unresectable MPM. All prior cytotoxic toxicities must have resolved to grade ≤ 1 prior to registration
* Measurable disease on CT scan, according to modified RECIST Criteria for Mesothelioma (Byrne MJ, 2004)
* Life expectancy ≥ 12 weeks
* Adequate hematologic and organ function, defined by the following laboratory results, obtained within 14 days prior to the first study treatment:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/µL (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1)
  * WBC count ≥ 3000 cells/µL
  * Lymphocyte count ≥ 250 cells/µL
  * Platelet count ≥ 100.000/µL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
  * Hemoglobin ≥ 5.6 mmol/L
  * Serum albumin ≥ 25 gr/L
  * AST, ALT and alkaline phosphatase ≤ 2.5 x ULN, with the following exceptions: patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN
  * Serum bilirubin ≤ 1.5 x ULN Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled
  * INR and aPTT ≤ 1.5 x ULN Patients receiving therapeutic anticoagulation should be on a stable dose Creatinine clearance ≥ 45 mL/min Cockcroft-Gault, Chronic Kidney Disease Epidemiology Collaboration or Modification of Diet in Renal Disease formulae may be used; 24-hour urine collection is not required
* Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus) and men with partners of childbearing potential, must agree to use adequate contraception (double barrier birth control) for the whole duration of study treatment and for 3 months after the last dose of therapy
* Women of childbearing potential must have a negative serum or urine pregnancy test within 48 hours prior the first dose of treatment

Exclusion Criteria:

* Medical or psychological impediment to comply with the protocol
* Patients with only peritoneal MPM
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, superficial or in-situ cancer of the bladder or other cancer for which the patient has been disease-free for at least five years
* Concomitant participation in another clinical trial (by the investigator's judgment)
* Uncontrolled pleural/peritoneal effusion, pericardial effusion or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled tumor-related pain Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions amenable to palliative radiotherapy should be treated prior to enrolment.
* Previous treatment with any checkpoint inhibitor
* Pregnant or lactating women
* Patients with brain metastases
* History of or active autoimmune disease (e.g. pneumonitis; rheumatoid arthritis; severe form of psoriasis; uncontrolled type I diabetes or hypothyroidism)
* History of idiopathic pulmonary fibrosis (including pneumonitis) or unresolved drug-induced pneumonitis, organizing pneumonia, or active pneumonitis on screening chest CT scan
* History of relevant gastrointestinal disease, including, but not limited to, Crohn's disease, ulcerative colitis, recurrent diverticulitis
* Prior allogenic bone marrow transplantation or prior solid organ transplantation
* History of HIV
* Patients with history of HBV infection are eligible if serological profile is compatible with past/resolved infection (defined as negative HBsAg test and positive antibody to HBV core antigen [anti-HBc] antibody test) and HBsAg test and HBV-DNA are both negative prior to Cycle 1, Day 1
* Patients with history of HCV infection must be screened for HCV-RNA PCR test prior to Cycle 1, Day 1, and are eligible if the test turns negative
* Other serious concomitant disease, including:

Active tuberculosis Severe infections within 4 weeks prior to Cycle 1, Day 1 Significant cardiovascular disease (NYHA class III or IV), myocardial infarction within the previous 6 months, unstable angina, or unstable arrhythmias Significant pulmonary (asthma or COPD) or hepatic disease or other illness considered by the investigator to constitute an unwarranted high risk for investigational treatment

* Major surgical procedures within 28 days prior to Cycle 1, Day 1
* Concurrent medications Treatment with systemic immunosuppressive medications, including but not limited to prednisone (with specific exceptions; see below), cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1.

The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.

The use of systemic prednisone at the dosage of 10 mg/day or lower (or equivalent) is allowed.

• Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Disease Controle Rate (DCR) at 12 weeks | at 12 weeks
  The number of patients that have CR or PR plus the number of patients with stable disease as a percentage of the total number of patients in the study.

SECONDARY OUTCOMES:
Safety: the incidence of adverse events, serious adverse events, deaths and laboratory abnormalities. | Participants will be followed for the duration of the trial, an expected average of 6 weeks
  Incidence of (serious) adverse events, serious adverse events, deaths and laboratory abnormalities.
Disease Controle Rate (DCR) at 6 months | at 6 months
  The number of patients that have CR or PR plus the number of patients with stable disease as a percentage of the total number of patients in the study.
Progression Free Survival (PFS) | Until progression, every 6 weeks up to 48 weeks
  The time from the date of start treatment to the date of the first documented tumor progression as determined by modified RECIST, or death due to any cause
Overall Survival (OS) | every 6 weeks up to 48 weeks, thereafter every 12 weeks up to 36 months.
  The time from date of start of treatment to the date of death from any cause, every 6 weeks up to 48 weeks, thereafter every 12 weeks up to 36 months
Overall Response Rate (ORR) | Every 6 weeks up to 48 weeks
  The number of subjects whose best confirmed objective response is a CR or PR, divided by the number of treated subjects

OTHER OUTCOMES:
Exploratory in blood and tumor biopsies | At screening and after 6 weeks of treatment (day 56-70)
  The research will focus on re-activation and expansion of tumor-specific T cells. Multimer pMCH technology will be used to examine the quantitative changes in T cell responses and transcriptomic analysis of tumor infiltrating T-cells in biopsies taken before and after 6 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Baas, MD, PhD, Principal Investigator — The Netherlands Cancer Institute-Antoni van Leeuwenhoek Ziekenhuis; Maria Disselhorst, MD, Principal Investigator — The Netherlands Cancer Institute-Antoni van Leeuwenhoek Ziekenhuis
Locations (1):
- Netherlands Cancer Institute-Antoni van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Desai AP, Kosari F, Disselhorst M, Yin J, Agahi A, Peikert T, Udell J, Johnson SH, Smadbeck J, Murphy S, Karagouga G, McCune A, Schaefer-Klein J, Borad MJ, Cheville J, Vasmatzis G, Baas P, Mansfield A. Dynamics and survival associations of T cell receptor clusters in patients with pleural mesothelioma treated with immunotherapy. J Immunother Cancer. 2023 Jun;11(6):e006035. doi: 10.1136/jitc-2022-006035. PMID 37279993
- [Derived] Mankor JM, Disselhorst MJ, Poncin M, Baas P, Aerts JGJV, Vroman H. Efficacy of nivolumab and ipilimumab in patients with malignant pleural mesothelioma is related to a subtype of effector memory cytotoxic T cells: Translational evidence from two clinical trials. EBioMedicine. 2020 Dec;62:103040. doi: 10.1016/j.ebiom.2020.103040. Epub 2020 Nov 7. PMID 33166791
- [Derived] Disselhorst MJ, Quispel-Janssen J, Lalezari F, Monkhorst K, de Vries JF, van der Noort V, Harms E, Burgers S, Baas P. Ipilimumab and nivolumab in the treatment of recurrent malignant pleural mesothelioma (INITIATE): results of a prospective, single-arm, phase 2 trial. Lancet Respir Med. 2019 Mar;7(3):260-270. doi: 10.1016/S2213-2600(18)30420-X. Epub 2019 Jan 16. PMID 30660511